CLINICAL TRIAL: NCT00717457
Title: Randomized, Active Controlled, Open Label Study to Compare Taspoglutide vs Exenatide as add-on Treatment to Metformin and/or Thiazolidinediones in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Taspoglutide Versus Exenatide for the Treatment of Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin, Thiazolidinedione or a Combination of Both.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC21625; 2008-001856-36
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; taspoglutide

ARMS (3):
- exenatide (Active Comparator)
  Interventions: Drug: exenatide
- taspoglutide 10mg (Experimental)
  Interventions: Drug: taspoglutide
- taspoglutide 10mg/20mg (Experimental)
  Interventions: Drug: taspoglutide

INTERVENTIONS:
Drug: exenatide — 5mg twice daily for 4 weeks followed by 10mg twice daily
  Arms: exenatide
Drug: taspoglutide — 10mg once weekly
  Arms: taspoglutide 10mg
Drug: taspoglutide — 10mg once weekly for 4 weeks followed by 20mg once weekly
  Arms: taspoglutide 10mg/20mg

SUMMARY:
This 3-arm study will assess the efficacy, safety and tolerability of taspoglutide compared with exenatide in patients with type 2 diabetes mellitus inadequately controlled with metformin, thiazolidinedione or a combination of both. Patients will be randomized to receive taspoglutide (10mg once weekly or 10mg once weekly for 4 weeks followed by 20mg once weekly) or exenatide (5 micrograms twice daily for 4 weeks followed by 10 micrograms twice daily) in a ratio of 1:1:1 in addition to continued prestudy metformin and thiazolidinedione either alone or in combination. The anticipated time on study treatment is 3+ years, and the target sample size is >500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes receiving metformin and/or pioglitazone or rosiglitazone for at least 12 weeks;
* HbA1c >=7.0% and <=10% at screening;
* BMI >=25kg/m2 (>23kg/m2 for Asians) and <=45kg/m2 at screening;
* stable weight +/- 5% for at least 12 weeks prior to screening.

Exclusion Criteria:

* history of type 1 diabetes, diabetes resulting from pancreatic injury or secondary forms of diabetes;
* history of acute metabolic diabetic complications within the previous 6 months;
* evidence of clinically significant diabetic complications;
* known proliferative diabetic retinopathy;
* myocardial infarction (MI), coronary artery bypass surgery, post-transplantation cardiomyopathy (PTCM) or stroke within the past 6 months;
* any abnormality in clinical laboratory test or ECG, which precludes safe involvement in the study as judged by the investigator;
* known hemoglobinopathy or chronic anemia;
* clinically significant gastrointestinal disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Fasting body weight | 24 weeks
Proportion of patients reaching target HbA1c <=7.0%, <=6.5% | 24 weeks
Relative change in glucose, insulin, C-peptide and glucagon values during a meal tolerance test in a subset of patients. | 24 weeks
Beta cell function (proinsulin/insulin ratio) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (183):
- United States (81):
  - Haleyville, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Tuscaloosa, Alabama
  - Little Rock, Arkansas
  - Escondido, California
  - La Jolla, California
  - Mission Viejo, California
  - Orange, California
  - Palm Springs, California
  - Rancho Cucamonga, California
  - Sacramento, California
  - San Leandro, California
  - Colorado Springs, Colorado
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Green Cove Springs, Florida
  - Jacksonville, Florida
  - Miami Beach, Florida
  - Niceville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Suwanee, Georgia
  - Chicago, Illinois
  - Lombard, Illinois
  - Peoria, Illinois
  - Evansville, Indiana
  - New Albany, Indiana
  - Iowa City, Iowa
  - Munfordville, Kentucky
  - Metairie, Louisiana
  - Bangor, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Rockville, Maryland
  - Royal Oak, Michigan
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Omaha, Nebraska
  - Concord, New Hampshire
  - Trenton, New Jersey
  - Voorhees Township, New Jersey
  - Whitehouse, New Jersey
  - Brooklyn, New York
  - New York, New York
  - Rochester, New York
  - Smithtown, New York
  - Springfield Gardens, New York
  - Staten Island, New York
  - Syracuse, New York
  - West Seneca, New York
  - Westfield, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Huntersville, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Westlake, Ohio
  - Medford, Oregon
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Red Lion, Pennsylvania
  - Providence, Rhode Island
  - Clemson, South Carolina
  - Columbia, South Carolina
  - Hickory Grove, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Everett, Washington
- Buenos Aires, Argentina
- Australia (2):
  - Camperdown, New South Wales
  - Freemantle, Queensland
- Brazil (6):
  - Goiânia, Goiás
  - Curtiba, Paraná
  - Belém, Pará
  - Porto Alegre, Rio Grande do Sul
  - Mogi Das Cruzes - Sp, São Paulo
  - São Paulo, São Paulo
- Canada (4):
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Pointe-Claire, Quebec
- Ballerup Municipality, Denmark
- Finland (4):
  - Helsinki
  - Kuopio
  - Oulu
  - Turku
- France (6):
  - Corbeil-Essonnes
  - Dommartin-lès-Toul
  - Montpellier
  - Narbonne
  - Paris
  - Salouël
- Germany (17):
  - Aschaffenburg
  - Berlin
  - Damme
  - Dresden
  - Essen
  - Falkensee
  - Hamburg
  - Ludwigshafen
  - Mainz
  - München
  - Münster
  - Neuwied
  - Nuremberg
  - Pirna
  - Rhaunen
  - Villingen-Schwenningen
  - Zwenkau
- Thessaloniki, Greece
- Guatemala City, Guatemala
- Israel (8):
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (5):
  - Pordenone, Friuli Venezia Giulia
  - Genoa, Liguria
  - Pavia, Lombardy
  - Olbia, Sardinia
  - Siena, Tuscany
- Mexico (7):
  - Acapulco
  - Aguascalientes
  - Chihuahua City
  - Durango
  - Guadalajara
  - Monterrey
  - Tampico
- Auckland, New Zealand
- Peru (2):
  - Arequipa
  - Lima
- Ponce, Puerto Rico
- Russia (11):
  - Barnaul
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - S. Petersburg
  - S.Petersburg
  - Saint Petersburg
  - Saratov
  - Tomsk
  - Yaroslavl
- South Africa (2):
  - Cape Town
  - Pretoria
- Seoul, South Korea
- Spain (4):
  - Bacarot Alicant, Alicante
  - Almería, Almeria
  - Madrid, Madrid
  - Alzira, Valencia
- Sweden (4):
  - Karlstad
  - Örebro
  - Stockholm
  - Uppsala
- Zurich, Switzerland
- Bangkok, Thailand
- Ukraine (6):
  - Dnipro
  - Donetsk
  - Kiev
  - Lviv
  - Odesa
  - Simferopol
- United Kingdom (5):
  - Bath
  - Bradford-on-Avon
  - Glasgow
  - Lanarkshire
  - Trowbridge

REFERENCES:
- [Derived] Rosenstock J, Balas B, Charbonnel B, Bolli GB, Boldrin M, Ratner R, Balena R; T-emerge 2 Study Group. The fate of taspoglutide, a weekly GLP-1 receptor agonist, versus twice-daily exenatide for type 2 diabetes: the T-emerge 2 trial. Diabetes Care. 2013 Mar;36(3):498-504. doi: 10.2337/dc12-0709. Epub 2012 Nov 8. PMID 23139373